CLINICAL TRIAL: NCT03095716
Title: Impact of Intraperitoneal Pressure and Warmed, Humidified CO2 Gas on Clinical Outcomes After Laparoscopic Surgery for Uterine Prolapse in Patients Aged ˃75 Years: A Observational Study
Brief Title: Laparoscopic Surgery in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-310
Record Dates: First submitted 2017-03-20; First posted 2017-03-30 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Uterine Prolapse
Keywords: Carbon dioxide pneumoperitoneum; Intraperitoneal pressure; Post-operative recovery; Laparoscopic Humidification System
MeSH Terms: conditions — Uterine Prolapse | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly patients: Impact of intraperitoneal pressure and warmed, humidified CO2 gas on clinical outcomes after laparoscopic surgery for uterine prolapse in patients aged ˃75 years
  Interventions: Other: laparoscopic surgery

INTERVENTIONS:
Other: laparoscopic surgery — Impact of intraperitoneal pressure and warmed, humidified CO2 gas on clinical outcomes after laparoscopic surgery for uterine prolapse in patients aged ˃75 years

SUMMARY:
The primary purpose is to evaluate the quality of post-operative recovery and post-operative pain in elderly patients (more than 75 years) who undergo laparoscopic surgery for uterine prolapse.

DETAILED DESCRIPTION:
Previous randomized clinical trial (NCT01887028) showed that the combined use of a low intraperitoneal pressure and a warmed, humidified CO2 gas resulted in better clinical outcomes (better quality of post-operative recovery and less post-operative pain) in patients aged 45-75 years, who underwent laparoscopic surgery for uterine prolapse.

Quality of post-operative recovery is very important in elderly patients. Investigators hypothesize that the combined use of a low intraperitoneal pressure and a warmed, humidified CO2 gas may also result in better clinical outcomes.

In this observational clinical trial, quality of post-operative recovery by QoR-40, post-operative pain by Visual Analog Scale, intra or postoperative complications and intraoperative core temperature are evaluated in elderly patients (more than 75 years old) who undergo laparoscopic surgery for uterine prolapse. Investigators use a low intraperitoneal pressure (6 mmHg) and a warmed, humidified CO2 gas during laparoscopy.

These outcomes will be compared with those of previous randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 75 years old
* Patients undergoing laparoscopic promontofixation with or without sub-total hysterectomy for uterine prolapse
* ASA class I or II

Exclusion Criteria:

* BMI more than 30
* Height less than 150cm

Min Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: ederly patients who undergo laparoscopic surgery for uterine prolapse
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Quality of post-operative recovery assessed by the Quality of Recovery-40 questionnaire | at 24h post-operatively
Quality of post-operative recovery assessed by the Quality of Recovery-40 questionnaire | at 48h post-operatively
Post-operative pain assessed by visual analogue scale in the postanesthesia care unit | at 24h post-operatively
Post-operative pain assessed by visual analogue scale in the word until discharge | at 24h post-operatively

SECONDARY OUTCOMES:
post operative complications | at 24h post-operatively
Intraoperative core temperature | at 24h post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Revaz Botchorishvili, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Matsuzaki S, Bonnin M, Fournet-Fayard A, Bazin JE, Botchorishvili R. Effects of Low Intraperitoneal Pressure on Quality of Postoperative Recovery after Laparoscopic Surgery for Genital Prolapse in Elderly Patients Aged 75 Years or Older. J Minim Invasive Gynecol. 2021 May;28(5):1072-1078.e3. doi: 10.1016/j.jmig.2020.09.017. Epub 2020 Sep 24. PMID 32979535